CLINICAL TRIAL: NCT00523419
Title: Phase II Trial of Pemetrexed in Second Line Advanced/Metastatic Osteosarcomas
Brief Title: Chemotherapy for Patients With Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11814; H3E-EW-S115 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Results first posted 2010-09-21 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed (Experimental): Participants received pemetrexed 500 milligrams per square meter (mg/m^2) by intravenous (IV) infusion of 10 minutes on Day 1 of each 21-day cycle.
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m^2, IV every 21 days until disease progression, unacceptable toxicity, participant or physician's decision.
  Other Names: LY231514; Alimta

SUMMARY:
The primary purpose of your participation in this study is to help answer the following research questions, and not to provide you treatment for your condition.

* To assess how well treatment with pemetrexed works for patients with your type of cancer
* To assess for any side effects that might be associated with pemetrexed.
* To look at the characteristics and levels of certain of your genes and proteins to learn more about osteosarcoma and how pemetrexed works in your body.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of high grade locally advanced or metastatic osteosarcoma
* Must have one prior chemotherapy regimen for advanced disease
* At least 1 unidimensional measurable lesion by computed tomography (CT) scan
* Have a good performance status
* Adequate organ function

Exclusion Criteria:

* Have a serious concomitant systemic disorder (for example active Human Immunodeficiency Virus infection)
* Have brain metastases not adequately treated
* Significant weight loss (that is more than 20%) over the previous 6 weeks before study entry
* Inability or unwillingness to take folic acid or vitamin B12 supplementation and corticosteroids
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villejuif
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newcastle upon Tyne, Tyneside, United Kingdom

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pemetrexed
Started | 32
Completed | 0
Not Completed | 32
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2
Not completed — Progressive Disease | 22
Not completed — Death due to Study Disease | 4
Not completed — Death due to Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed
Number analyzed (Participants) | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 42.1 (16.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 20
Region of Enrollment [Number; unit: participants]
  France | 13
  Spain | 3
  Germany | 6
  United Kingdom | 1
  Italy | 9
Best Response of Last Prior Treatment Regimen for Osteosarcoma [Number; unit: participants] — Complete response (CR): all tumor lesions disappear. Partial response (PR): >=30% decrease in sum of the longest diameter (LD) of target lesions (reference: baseline sum LDs) or complete disappearance of target lesions, with persistence (but not worsening) of >=1 nontarget lesions; no appearance of new lesions. Stable disease: neither sufficient shrinkage for PR nor sufficient increase for PD; references: smallest sum LD. Progressive disease (PD): >=20% increase in the sum of LD of target lesions (references: smallest sum LD recorded since treatment started) or appearance of >=1 new lesions.
  participants
    Complete Response | 1
    Partial Response | 3
    Stable Disease | 10
    Progressive Disease | 15
    Not Applicable | 3
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — 0: fully active, able to carry on all pre-disease performance without restriction; 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2: ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours; 3: capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4: completely disabled, cannot carry on any self-care, totally confined to bed or chair; 5: dead.
  participants
    ECOG Performance Status 0 | 16
    ECOG Performance Status 1 | 14
    ECOG Performance Status 2 | 1
    ECOG Performance Status Not Available | 1
Histopathological Diagnosis of Osteosarcoma at Study Entry [Number; unit: participants] | 32
Number of Target Lesions [Number; unit: participants] — Target lesions: all measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs; selected on the basis of size (those lesions with the longest diameter) and suitability for accurate repeated measurements (either by imaging techniques or clinically). If the measurable disease is restricted to a solitary lesion, the neoplastic nature of the lesion was confirmed by cytology/histology.
  participants
    0 Target Lesions | 1
    1 Target Lesion | 9
    2 Target Lesions | 8
    3 Target Lesions | 4
    4 Target Lesions | 3
    5 Target Lesions | 7
Number of non target lesions [Number; unit: participants] — All lesions that do not meet the criteria for target lesions, including small lesions (longest diameter <20 millimeter [mm] with conventional computed tomography [CT] scan, <10 mm with spiral CT scan) and other non-measurable lesions.
  participants
    0 Non Target Lesions | 10
    1 Non Target Lesion | 15
    2 Non Target Lesions | 5
    3 Non Target Lesions | 1
    5 Non Target Lesions | 1
Pathological Diagnosis of Osteosarcoma at Study Entry [Number; unit: participants] | 32
Time from last diagnosis to enrollment [Mean (Standard Deviation); unit: days] | 13.3 (12.10)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Tumor Response
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR) = disappearance of all target lesions; Partial Response (PR) = at least a 30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD) = at least a 20% increase in sum of longest diameter of target lesions; Stable Disease (SD) = small changes that do not meet above criteria. Tumor Response Rate(%) = sum of number of PR + CR observed/number of participants qualified for tumor response analysis * 100.
Time Frame: Baseline to 21 months
Population: Participants who qualified for tumor response analysis are those with histological evidence of high grade locally advanced or metastatic osteosarcoma and treatment with at least 1 dose of study drug. Three participants died before the first tumor assessment and 1 participant discontinued without any tumor assessments and were considered Unknown.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 32
percentage of participants
  Response Rate | 3.1 [0.1 to 16.2]
  Complete Response (CR) | 0 [0 to 0]
  Partial Response (PR) | 3.1 [0.1 to 16.2]
  Stable Disease (SD) | 15.6 [5.3 to 32.8]
  Progressive Disease (PD) | 68.8 [50.0 to 83.9]
  Unknown | 12.5 [3.5 to 29.0]

2. Secondary Outcome: Time to Treatment Failure
Description: When the protocol was written, time to treatment failure (TTTF) was included as a secondary endpoint. However, it was subsequently realized that due to the design of the study, participants are treated until disease progression or discontinuation from study treatment, not for a fixed number of cycles. Therefore, it was concluded that analysis of TTTF was inappropriate with the current study design and the analysis was not conducted, since it would be essentially the same as Progression-Free Survival.
Time Frame: Baseline to 21 months
Population: Since this outcome measure was not analyzed due to the study design, zero participants were analyzed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pemetrexed
Number analyzed (Participants) | 0

3. Secondary Outcome: Correlation of Disease Outcome With Pharmacogenomic Analysis
Description: It was planned to examine methylthioadenosine phosphorylase (MTAP) gene deletion, folate receptor alpha (FRα) and folylpoly-gamma-glutamate synthetase (FPGS) expression, and to correlate the results with the clinical data to determine the association between these factors and clinical outcome to treatment. However, due to the small number of participants with partial response (n=1), the planned statistical analyses that would correlate responders/non responders with pharmacogenomics data are no longer valid and the analyses were not conducted.
Time Frame: Baseline to 21 months
Population: Since this outcome measure was not analyzed due to the inadequate number of responders, zero participants were analyzed.
Measure: Number; unit: correlation coefficient
Arm/Group | Pemetrexed
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Adverse Events (Pharmacology Toxicity)
Description: Pharmacology toxicity was defined as serious and non-serious adverse events. Summaries of these adverse events are located in the Reported Adverse Event Section.
Time Frame: Baseline to 21 months
Population: Full analysis population: all participants who were treated with at least one dose of the study regimen
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 32
participants
  Serious Adverse Events | 11
  All Other Nonserious Adverse Events | 26

5. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from the first objective status assessment of CR or PR to the first date of progression or death as a result of any cause: CR was achieved if all tumor lesions disappeared; PR was achieved if there was >=30% decrease in sum of the longest diameter (LD) of target lesions (reference: baseline sum LDs) or complete disappearance of target lesions with persistence (but not worsening) of >=1 nontarget lesions and no appearance of new lesions.
Time Frame: Baseline to 31 months
Population: Tumor response population: participants with best overall response of complete response (CR) and partial response (PR).
Measure: Number; unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 1
months | 9.5 [4.0 to NA]

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was from date of study enrollment to first date of objectively determined progressive disease (PD) or death from any cause. For participants who did not die as of data cut-off date and who did not have objective PD, PFS was censored at date of last objective progression-free disease assessment. For participants who received subsequent systemic anticancer therapy (after discontinuation from study drug) before objectively determined disease progression or death, PFS was censored at date of last objective progression-free disease assessment, before post-discontinuation chemotherapy.
Time Frame: Baseline to 10.4 months
Population: Full analysis population: all participants who were treated with at least one dose of the study regimen.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 32
months | 1.4 [1.4 to 1.7]

7. Secondary Outcome: Overall Survival (OS) Time
Description: OS was the duration from enrollment to death. For participants who lived, OS was censored at the last contact.
Time Frame: Baseline to 27.6 months
Population: Full analysis population: all participants who were treated with at least one dose of the study regimen.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 32
months | 5.5 [2.3 to 10.5]

ADVERSE EVENTS:
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 11/32
Other Adverse Events (participants affected / at risk) | 26/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=32)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) — Resulted in death due to multiorgan failure possibly related to study drug.
Pyrexia (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1) — Cause of death could not be established.
Catheter related infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vertebroplasty (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=32)
Anaemia (Blood and lymphatic system disorders) | 6 (7)
Leukopenia (Blood and lymphatic system disorders) | 3 (5)
Neutropenia (Blood and lymphatic system disorders) | 3 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 2 (9)
Nausea (Gastrointestinal disorders) | 4 (14)
Vomiting (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 8 (14)
Fatigue (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 4 (4)
Pain (General disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (5)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Dizziness (Nervous system disorders) | 2 (10)
Headache (Nervous system disorders) | 2 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 4 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days